CLINICAL TRIAL: NCT04891328
Title: The Experience of Participating in a Pediatric Summer Intensive Therapy Program--A Mixed Methods Study
Brief Title: Experience With a Pediatric Summer Intensive Therapy Program
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jamie Hall, Assistant Teaching Professor, University of Missouri-Columbia
Other Study IDs: 2058022
Record Dates: First submitted 2021-04-29; First posted 2021-05-18 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Neurodevelopmental Disorders
Keywords: pediatric rehabilitation; intensive therapy
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Intensive therapy program — The intensive therapy program consists of physical therapy, occupational therapy, and speech therapy 3-6 hours x 4-5 days/week for 4 weeks. The individual therapies received will vary with the child/caregiver goals and be based on neuroplasticity and motor learning principles.

SUMMARY:
The purpose of this study is to explore the lived experiences of children with neurodevelopmental diagnoses and their caregivers with an intensive model of therapy. Children will receive usual care during the summer intensive program and the investigators will access medical records to assess effectiveness. Children and caregivers will also be asked to participate in semi-structured interviews upon the completion of the episode of care.

DETAILED DESCRIPTION:
The purpose of this study is to explore the lived experiences of children with neurodevelopmental diagnoses and their caregivers with an intensive model of therapy. Research questions include: 1.) What are the perceptions of children and caregivers about intensive therapy after participating in multiple intensive therapy episodes over time? 2.) Why do caregivers choose to continue with an intensive model of therapy periodically for their child with neurodevelopmental diagnoses? 3.) What were the outcomes for children with neurodevelopmental disabilities participating in an episode of intensive therapy? Children will receive usual care during the summer intensive program and the investigators will access medical records to assess effectiveness. Children and caregivers will also be asked to participate in semi-structured interviews upon the completion of the episode of care.

ELIGIBILITY:
Inclusion Criteria:

* Children receiving therapy through the Children's Therapy Center's Tiger Intensive Program and their caregivers from May 24 to August 13 2021.

Exclusion Criteria:

* n/a

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 4-15 years old with neurodevelopmental diagnoses and scheduled for an intensive therapy program over the summer.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Semi-structured interviews | at discharge assessed up to 10 days
  Upon completion of the program, children and caregivers will participate in an interview about their experience
Canadian Occupational Performance Measure | measured at discharge 4 weeks after enrollment
  Individualized client-centered performance measure

SECONDARY OUTCOMES:
Change in Lower extremity passive range of motion | Measured at day 1 and discharge 4 weeks later
  Measured at ankle, knee, and hip with goniometer
Change in Thomas Test | Measured at day 1 and discharge 4 weeks later
  Hip flexor length test
Change in popliteal angle | Measured at day 1 and discharge 4 weeks later
  Hamstring length test
Change in Gastrocnemius muscle length | Measured at day 1 and discharge 4 weeks later
  Measured with goniometer
Change in Kids Bestest | Measured at day 1 and discharge 4 weeks later
  Balance measure for pediatric patients
Change in m-CTSIB | Measured at day 1 and discharge 4 weeks later
  Balance measure
Change in Early Clinical Assessment of Balance | Measured at day 1 and discharge 4 weeks later
  Balance measure
Change in Segmental Assessment of Trunk Control (SATCO) | Measured at day 1 and discharge 4 weeks later
  Measurement of trunk control
Change in Edinburgh Visual Gait Scale | Measured at day 1 and discharge 4 weeks later
  Observational Gait measure
Change in Timed Up and Down Stairs | Measured at day 1 and discharge 4 weeks later
  Measure of stair performance
Change in Timed on and off the floor | Measured at day 1 and discharge 4 weeks later
  Measure of transition from floor to standing
Change in 6 minute walk test | Measured at day 1 and discharge 4 weeks later
  Measure of walking performance
Change in Peds QL | Measured at day 1 and discharge 4 weeks later
  Pediatric quality of life measure
Change in GOAL | Measured at day 1 and discharge 4 weeks later
  patient reported measure of function mobility
Change in Pediatric Evaluation of Disability Inventory | Measured at day 1 and discharge 4 weeks later
  Measure of amount of disability
Pediatric Balance Scale | Measured at day 1 and discharge 4 weeks later
  Measure of balance

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri Healthcare Children's Therapy Center, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No